CLINICAL TRIAL: NCT02959476
Title: A Double Blind, Multi-center, Randomized, Placebo-Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Ropivacaine 0.2% Pre-Filled Dispenser for the Treatment of Postsurgical Pain in Patients Undergoing Cesarean Delivery
Brief Title: Ropivacaine 0.2% Pre-Filled Dispenser for the Treatment of Postsurgical Pain in Patients Undergoing Cesarean Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioQ Pharma, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 94006184
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; Postsurgical pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ropivacaine 0.2% (Experimental): Naropin® (ropivacaine HCl Injection, USP) bolus + Ropivacaine 0.2% Pre-Filled Dispenser infusion - "Ropivacaine Infusion treatment arm"
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Naropin® (ropivacaine HCl Injection, USP) bolus + placebo infusion (normal saline) - "Placebo treatment arm"
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ropivacaine — Anesthetic
  Arms: Ropivacaine 0.2%
Drug: Placebos — Inactive comparator
  Arms: Placebo

SUMMARY:
This study evaluates a Ropivacaine 0.2% Pre-Filled Dispenser in the treatment of post-surgical pain in patients undergoing Cesarean delivery. Half of the patients will receive Ropivicaine and half will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Complete the informed consent process as documented by a signed informed consent form (ICF).
* Be in generally good health and classified as either PS-1 or PS-2 by the American Society of Anesthetists (ASA) Physical Status Classification System.
* Have a single birth pregnancy. Can be parous or nulliparous.
* Be scheduled for a Cesarean Delivery
* Subjects undergoing emergency Cesarean Delivery will not be eligible for participation in this study.
* In the event a subject signs the ICF (but has not been randomized), has a C section planned and then has an emergency C section delivery, this subject will be considered a screen failure.
* In the unlikely event a subject signs the ICF and is randomized into the study, has a C section planned and then has an emergency C section delivery, this subject will continue in the study as planned.
* Be willing to complete the pain assessments according to the protocol and return to clinic as scheduled, as needed.

Exclusion Criteria:

* Have an uncontrolled medical condition, serious intercurrent illness, clinically significant general health condition, or extenuating circumstance that may significantly decrease study compliance or otherwise preclude their participation in the study.
* Have a clinically significant abnormal electrocardiogram (ECG) at screening as determined by the Investigator.
* Have a history of any medical condition or surgical procedure that would alter the absorption, distribution, metabolism, or excretion of ropivacaine.
* Have, in the opinion of the investigator, a clinically significant abnormality in their clinical laboratory values (urinalysis, hematology and chemistry) at screening.
* Have made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 56 days prior to Day 1.
* Weigh greater than 100 kg (220 lbs).
* Have made a plasma donation within 7 days prior to Day -1.
* Have a known allergy or hypersensitivity to anesthetics (eg. Ropivacaine), acetaminophen, or non-steroidal anti inflammatory drugs (NSAIDs, eg, ibuprofen or naproxen, ketorolac).
* Not be able or willing to discontinue the prohibited medications listed below within the allotted time before surgery and throughout the duration of their participation in the study.

  * monoamine oxidase inhibitors (MAOIs) within the past 30 days
  * anticonvulsants, tricyclic antidepressants (TCAs), neuroleptics, serotonin-norepinephrine reuptake inhibitors (SNRIs), as well as selective serotonin reuptake inhibitors (SSRIs) (unless SSRIs have been prescribed for depression and/or anxiety and subjects have been on a stable dose for at least 30 days prior to the screening visit);
  * Corticosteroids: Oral and injectable corticosteroids must be discontinued 3 months prior to surgery; nasal, inhaled and topical corticosteroids will be allowed;
* Use concurrent therapy that could interfere with the evaluation of efficacy or safety parameters in the opinion of the investigator (eg, any drugs, in the investigator's opinion, that may exert significant analgesic properties), except for rescue medications.
* Have a history of seizures or history of serious head injury.
* Must not be a member of a vulnerable population as defined by the Code of Federal Regulations Title 45, Part 46, Delivery 46.111(b), including but not limited to employees (temporary, part-time, full-time, etc.) or a family member of the research staff conducting the study, or of the Sponsor, or of the Clinical Research Organization.
* Have previously participated in a clinical trial using ropivacaine.
* Have a history of major mental illness that in the opinion of the Investigator may affect the ability of the subject to participate in the study. Institutionalized subjects will not be eligible for participation.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Cumulative analgesic effect | 48 hours

SECONDARY OUTCOMES:
Use of other analgesics | 48 hours
Local safety and tolerability using descriptive statistics of the evaluation of physical exams, wound healing and treatment-emergent adverse events local to the surgical wound | 7 days
Overall safety using descriptive statistics of the evaluation of physical exam, vital signs, clinical laboratory tests, and treatment-emergent adverse events | 7 days
Analgesic effect at specified intervals | 48 hours

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Clinical Research Associates, Inc., Birmingham, Alabama
  - Shoals Medical Trials, Inc., Sheffield, Alabama
  - University of California, Irvine, Orange, California
  - Vision Clinical Research, Wellington, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - MedPharmics, LLC, Biloxi, Mississippi
  - Duke University Medical Center, Durham, North Carolina
  - Compass Clinical Trial, Beaumont, Texas
  - Physician's Research Options, LLC- Corner Canyon OB/GYN, Draper, Utah
  - Health Sciences Center- University of Utah, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia